CLINICAL TRIAL: NCT06031818
Title: Usability and Clinical Effectiveness of an Interpretable Deep Learning Framework (VAE-MILP) Using Counterfactual Explanations and Layerwise Relevance Propagation Framework for Post-Hepatectomy Liver Failure Prediction
Brief Title: Usability and Clinical Effectiveness of an Interpretable Deep Learning Framework for Post-Hepatectomy Liver Failure Prediction
Status: Recruiting | Type: Observational
Sponsor: Maastricht University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: Interpretable DL; 92059201 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Post-hepatectomy Liver Failure; Hepatocellular Carcinoma; Artificial Intelligence
Keywords: deep learning; interpretability; post-hepatectomy liver failure; hepatocellular carcinoma; shear wave elastography
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HCC: Patients who underwent curative liver resection for HCC in the First Affiliated Hospital of Sun Yat-Sen University in China.
  Interventions: Other: The explanation of deep learning framework (VAE-MLP) , including counterfactual explanations and layerwise relevance propagation; Other: The model prediction; Other: The model prediction and the explanation of deep learning framework (VAE-MLP) , including counterfactual explanations and layerwise relevance propagation

INTERVENTIONS:
Other: The explanation of deep learning framework (VAE-MLP) , including counterfactual explanations and layerwise relevance propagation — The radiologist and clinicians will be provided the model prediction results with the explanation of the model and they will fill in a questionnaire to evaluate the usability of the interpretable framework.
Other: The model prediction — The radiologist and clinicians will be provided the model prediction results without the explanation of the model and they will be asked to give their own prediction.
Other: The model prediction and the explanation of deep learning framework (VAE-MLP) , including counterfactual explanations and layerwise relevance propagation — The radiologist and clinicians will be provided the model prediction results with the explanation of the model and they will be asked to give their own prediction.

SUMMARY:
The goal of this in-silico clinical trial is to learn about the usability and clinical effectiveness of an interpretable deep learning framework (VAE-MLP) using counterfactual explanations and layerwise relevance propagation for prediction of post-hepatectomy liver failure (PHLF) in patients with hepatocellular carcinoma (HCC). The main questions it aims to answer are:

* To investigate the usability of the VAE-MLP framework for explanation of the deep learning model.
* To investigate the clinical effectiveness of VAE-MLP framework for prediction of post-hepatectomy liver failure in patients with hepatocellular carcinoma.

In the usability trial the clinicians and radiologists will be shown the counterfactual explanations and layerwise relevance propagation (LRP) plots to evaluate the usability of the framework.

In the clinical trial the clinicians and radiologists will make the prediction under two different conditions: with model explanation and without model explanation with a washout period of at least 14 days to evaluate the clinical effectiveness of the explanation framework.

DETAILED DESCRIPTION:
Post-hepatectomy liver failure (PHLF) is a severe complication after liver resection. It is important to develop an interpretable model for predicting PHLF in order to facilitate effective collaboration with clinicians for decision-making. Two-dimensional shear wave elastography (2D-SWE) is a liver stiffness measurement (LSM) technology that was proven to be useful in liver fibrosis staging. Therefore 2D-SWE shows the potential value for liver function assessment and PHLF prediction. 2D-SWE images display color-coded tissue stiffness map of liver parenchyma, with red representing a solid tissue (higher stiffness) and blue representing a soft tissue (lower stiffness). Routine analysis of 2D-SWE fails to fully utilize all information available in the images and also suffers from inter-observer variance in choosing the optimal quantification region.

Deep learning (DL) has demonstrated state-of-the-art performance on many medical imaging tasks such as classification or segmentation. However, despite significant progress in DL, the clinical translation of DL tools has so far been limited, partially due to a lack of interpretability of models, the so-called "black box" problem. Interpretability of DL systems is important for fostering clinical trust as well as timely correcting any faulty processes in the algorithms.

Here, the investigators present a novel interpretable DL framework (VAE-MLP) which incorporates counterfactual analysis for the explanation of 2D medical images and LRP for the explanation of feature attributions of both medical images and clinical variables.

The goal of this in-silico clinical trial is to learn about the usability and clinical effectiveness of an interpretable deep learning framework (VAE-MLP) using counterfactual explanations and layerwise relevance propagation for prediction of post-hepatectomy liver failure (PHLF) in patients with hepatocellular carcinoma. The main questions it aims to answer are:

* To investigate the usability of the the interpretable deep learning framework (VAE-MLP) for explanation of the deep learning model.
* To investigate the clinical effectiveness of the interpretable deep learning framework (VAE-MLP) for prediction of post-hepatectomy liver failure in patients with hepatocellular carcinoma.

In the usability trial the clinicians and radiologists will be shown the counterfactual explanations and layerwise relevance propagation plots of 6 examples. The score of the Likert scale of a designed questionnaire is used to evaluate the usability of the framework.

In the clinical trial the clinicians and radiologists will make the prediction under two different conditions: with model explanation and without model explanation with a washout period of at least 14 days. The accuracy, sensitivity and specificity is used to compare the clinical effectiveness of the explanation framework.

ELIGIBILITY:
Inclusion Criteria:

1. patients with treatment-naive and resectable HCC;
2. performance status Eastern Cooperative Oncology Group (PS) score 0-1.

Exclusion Criteria:

1. liver resection was not performed;
2. pathological diagnosis of non-HCC;
3. failure in liver stiffness measurement defined as the elastography color map was less than 75% filled or interquartile range (IQR)/median > 30%;
4. immune-active chronic hepatitis indicated by an elevation of alanine aminotransferase (ALT) levels ≥ 2×upper limit of normal (ULN);
5. obstructive jaundice or dilated intrahepatic bile ducts with a diameter of >3 mm;
6. hypoalbuminemia, hyperbilirubinemia, or coagulopathy not related to the liver.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent curative liver resection for HCC.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Clinical effectiveness of the explanation framework | From enrollment to the end of trial at 8 weeks
  The accuracy, sensitivity and specificity will be compared between the prediction made with and without the explanation of the DL model to determine the clinical effectiveness of the explanation framework.

SECONDARY OUTCOMES:
Usability of the explanation framework | From enrollment to the end of trial at 8 weeks
  The score of the Likert scale of a designed questionnaire is used to evaluate the usability of the framework. Each item is given a score from 1 to 5. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, Principal Investigator — Maastricht University
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) can be shared if asked